CLINICAL TRIAL: NCT02236520
Title: Tissue Sodium in Pre-hypertensive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 141382
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-04

CONDITIONS: Hypertension
Keywords: Na+ MRI; salt stores
MeSH Terms: conditions — Hypertension | interventions — Spironolactone; Chlorthalidone; Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Spironolactone (Active Comparator): 50 mg capsule of Spironolactone administered orally 1 per day for 8 weeks
  Interventions: Drug: Spironolactone
- Chlorthalidone (Active Comparator): 25 mg capsule of Chlorthalidone administered orally 1 per day for 8 weeks
  Interventions: Drug: Chlorthalidone
- Diet (Active Comparator): diet of 6 g salt per day for 8 weeks
  Interventions: Dietary Supplement: Diet
- Placebo (Placebo Comparator): placebo capsule administered orally 1 per day for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone
  Arms: Spironolactone
Drug: Chlorthalidone
  Arms: Chlorthalidone
Dietary Supplement: Diet
  Arms: Diet
Drug: Placebo
  Arms: Placebo

SUMMARY:
Cardiovascular disease is the first common cause of death worldwide. Hypertension is the number one driving risk factor. Hypertension has long been associated with dietary salt intake. We believe that the accumulation of salt in the interstitium and inside cells represents a neglected risk factor, which initiates a pro-inflammatory state, chronically increases blood pressure, and leads to systemic energy imbalance. We will explore the concept that Na+ storage in the skin and in muscle is associated with increased blood pressure, a pro-inflammatory state, and reduced insulin sensitivity. We will do so by addressing the following specific aims:

* Specific Aim 1: To test the hypothesis that African Americans are characterized by increased tissue Na+ storage, which is paralleled by higher blood pressure, reduced forearm blood flow, and enhanced pulse wave velocity
* Specific Aim 2: To test the hypothesis that treatment with spironolactone reduces tissue Na+ content
* Specific Aim 3: To test the hypothesis that Na+ storage leads to immune cell activation
* Specific Aim 4: To test the hypothesis that the accumulation of salt in skin and muscle is associated with decreased insulin sensitivity and propensity to diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 80 years old;
* Systolic blood pressures between 110 to 150 mmHg and/or diastolic blood pressure between 80-99 mmHg;
* Ability to give informed consent.

Exclusion Criteria:

* Pregnancy;
* Intolerance to study protocols;
* Acute cardiovascular events within the previous 6 months;
* Impaired renal function [estimated glomerular filtration rate (GFR) < 45 ml/min/1.73m^2];
* Current or recent treatment with systemic glucocorticoid therapy (within 1 month of enrollment);
* Current use of anti-hypertensive medication (except calcium channel blockers and beta blockers);
* Diabetes mellitus requiring medical therapy;
* Morbid obesity (BMI > 45);
* Prior adverse reaction to a thiazide or spironolactone;
* Claustrophobia preventing the patient from having an MRI or other contraindications to MRI;
* Impaired hepatic function (aspartate amino transaminase and/or alanine amino transaminase > 1.5x upper limit of normal range);
* Current illicit drug use;
* Sexually active women of childbearing potential** who are unwilling to practice adequate contraception during the study [adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device (IUD); bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly].

  * Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University; Jens Titze, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Ertuglu LA, Sahinoz M, Alsouqi A, Deger SM, Guide A, Stewart TG, Pike M, Robinson-Cohen C, Akwo E, Pridmore M, Crescenzi R, Madhur MS, Harrison DG, Luft FC, Titze J, Ikizler TA. High tissue-sodium associates with systemic inflammation and insulin resistance in obese individuals. Nutr Metab Cardiovasc Dis. 2023 Jul;33(7):1398-1406. doi: 10.1016/j.numecd.2023.03.024. Epub 2023 Apr 10. PMID 37156670
- [Derived] Alsouqi A, Deger SM, Sahinoz M, Mambungu C, Clagett AR, Bian A, Guide A, Stewart TG, Pike M, Robinson-Cohen C, Crescenzi R, Madhur MS, Harrison DG, Ikizler TA. Tissue Sodium in Patients With Early Stage Hypertension: A Randomized Controlled Trial. J Am Heart Assoc. 2022 Apr 19;11(8):e022723. doi: 10.1161/JAHA.121.022723. Epub 2022 Apr 18. PMID 35435017

RESULTS

PARTICIPANT FLOW:
Groups:
- Spironolactone: 50 mg capsule of Spironolactone administered orally 1 per day for 8 weeks
  Spironolactone
- Chlorthalidone: 25 mg capsule of Chlorthalidone administered orally 1 per day for 8 weeks
  Chlorthalidone
- Diet: diet of 6 g salt per day for 8 weeks
  Diet
- Placebo: placebo capsule administered orally 1 per day for 8 weeks
  Placebo
Period: Overall Study
Arm/Group | Spironolactone | Chlorthalidone | Diet | Placebo
Started | 16 | 13 | 15 | 15
Completed | 14 | 8 | 15 | 14
Not Completed | 2 | 5 | 0 | 1
Not completed — Physician Decision | 0 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Chlorthalidone | Diet | Placebo | Total
Number analyzed (Participants) | 16 | 13 | 15 | 15 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (11) | 49 (9) | 49 (13) | 48 (14) | 48 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 9 | 10 | 40
  Male | 5 | 3 | 6 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 15 | 13 | 15 | 15 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 5 | 8 | 6 | 26
  White | 9 | 8 | 7 | 9 | 33
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 15 | 15 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Tissue Sodium Concentration Measured Using Sodium Magnetic Resonance Imaging (NaMRI)
Description: NaMRI is a sensitive laboratory assessment of the concentration of sodium in tissue
Time Frame: baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Spironolactone | Chlorthalidone | Diet | Placebo
Number analyzed (Participants) | 14 | 8 | 15 | 14
mmol/L | -0.202 [-0.973 to 1.667] | 0.430 [-1.085 to 1.285] | -1.745 [-2.157 to -0.219] | -0.407 [-2.108 to 1.088]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Spironolactone | Chlorthalidone | Diet | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/16 | 2/13 | 1/15 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spironolactone (N=16) | Chlorthalidone (N=13) | Diet (N=15) | Placebo (N=15)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gastrointestinal upset (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02236520/Prot_SAP_000.pdf